CLINICAL TRIAL: NCT05163340
Title: Nurses' Views on Alarm Fatigue and Its Reduction in Adult Intensive Care Units: Convergent Parallel Design
Brief Title: Views of Nurses on Alarm Fatigue in ICUs
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Fatma CEBECİ, Fatma CEBECİ, Akdeniz University
Other Study IDs: KAEK-271
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Nurse's Role
Keywords: Alarm fatigue; Intensive care; Nursing; Mixed method
MeSH Terms: conditions — Alert Fatigue, Health Personnel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study focused on determining the views of nurses on alarm fatigue and its reduction in adult intensive care units.

DETAILED DESCRIPTION:
Backround: Physiological monitoring of critically ill patients in ICU is a complex nursing task, and nurses are key professionals managing multiple monitoring devices.

Aim: The aim of this study is to determine the views of nurses on alarm fatigue and its prevention in adult intensive care units.

Study Design: In the study, the minimum sample size was calculated as 67 for a population size of 106 and a 95% confidence interval, taking into account the alarm fatigue standard deviation (σ=6.82) found in the Turkish validity study of the "Nurses' Alarm Fatigue Scale" (t=1.96; d=1) . Considering that there may be losses, 74 nurses will be included in the study by taking 10% more. In the qualitative phase of the research, intensive care nurses who agreed to be interviewed during the collection of quantitative data will be included.

Method: In this study, parallel data type will be used in convergent parallel mixed design. The quantitative phase of the study is a descriptive study to determine alarm fatigue levels in nurses working in adult intensive care units. In the qualitative phase of the research; A case study will be conducted at the same time in order to examine the findings revealed with quantitative data in more depth and to determine the views of nurses on reducing alarm fatigue. Individual in-depth interviews will be held in a suitable room using the "Semi-Structured Interview Form" created by the researchers with those who agree to participate in the qualitative study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Who volunteered to participate in the research
* Working in adult intensive care units

Exclusion Criteria:

* Under the age of 18
* Not working in adult intensive care unit

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The research populations consists of nurses working in adult ICU a University Hospital. The sample number was calculated with the formula known population and the cases average of the event in the study. In this study, considering the alarm fatigue standard deviation (σ=6.82) found in the Turkish validity study of the scale, the minimum sample size was calculated as 67 for a population size of 106 and a 95% confidence interval (t=1.96; d=1). Considering that there may be losses 10% more (74 nurses) will be taken.
  The qualitative phase of the research will be with nurses who agreed to be interview and will be terminated when the data reach the saturation point and no new information emerge.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Nurses' Alarm Fatigue Scale | 30 May 2022
  The scale consists of 9 items and the score range is between 0-36. High scores indicate the effects of alarm fatigue on nurses' performance. Each item in the questionnaire is scored between 0 and 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

REFERENCES:
- [Derived] Ucak A, Cebeci F, Tat Catal A. Nurses' Alarm Fatigue Levels in Adult Intensive Care Units and Their Strategies to Reduce Fatigue: A Convergent Parallel Design. J Clin Nurs. 2025 May;34(5):1691-1703. doi: 10.1111/jocn.17644. Epub 2025 Jan 20. PMID 39831580